CLINICAL TRIAL: NCT03967574
Title: Characterization and Temporal Evaluation of the Effects of Subacromial Corticosteroid Injections and Trans-cranial Direct Current Stimulation in Rotator Cuff Tendinopathy
Brief Title: Subacromial Corticosteroid Injections and tDCS in Rotator Cuff Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Principal Investigator, Samuel Larrivée, Principal Investigator, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-158
Record Dates: First submitted 2019-05-26; First posted 2019-05-30 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Rotator Cuff Tendinosis; Rotator Cuff Impingement Syndrome; Rotator Cuff Impingement; Rotator Cuff Injuries; Rotator Cuff Syndrome of Shoulder and Allied Disorders
Keywords: transcranial direct current stimulation; non invasive brain stimulation; tDCS; NIBS; subacromial corticosteroid injection
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Impingement Syndrome | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: All participants received a subacromial corticosteroid injection.
  Two weeks following the injection, participants were randomized into 3 groups:
  * Anodal transcranial direct current stimulation (treatment group)
  * Placebo tDCS (placebo group)
  * No further intervention (control group)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and assessors were blind to the assignment of the treatment vs placebo group, while there was no feasible way to conceal the control group.
  Participants from the treatment and placebo group received the tDCS intervention by a care provider not involved in the recruitment, data collection or outcome assessment. The tDCS apparatus was out of sight of the participant for the duration of the treatment. Treatment patients received tDCS treatment for the whole duration of the planned intervention (20 minutes), while the device was only turned on for 30 seconds, then gradually turned off for the participants in the placebo group. This was done in order to mimic the initial sensation of tingling felt by participants in the treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Real tDCS (Experimental): Participants received the full tDCS intervention for a total of 20 minutes, one time, two weeks following the CSI
  Interventions: Device: Transcranial direct current stimulation
- Sham tDCS (Sham Comparator): The patients were set up in an identical way as with the real tDCS group, but only received active stimulation for 30 seconds, after which the current was gradually stopped. The participants continued wearing the electrodes until the end of the 20 minutes treatment.
  Interventions: Device: Transcranial direct current stimulation
- Control (No Intervention): Participants received no further intervention two weeks following their CSI

INTERVENTIONS:
Device: Transcranial direct current stimulation — The tDCS anode was applied on the primary motor cortex area responsible for the control of the rotator cuff, as determined using transcranial magnetic stimulation and surface electromyography. The cathode was applied on the contralateral forehead, just above the eyebrow. The electrodes were soaked in saline solution to improve conductivity and the montage was secured with rubber bands and adhesive tape.
  The tDCS device (Soterix Medical 1x1 tDCS device) was then gradually turned to an intensity of 2mA. This stimulation was continued for a total of 20 minutes, after which it was gradually stopped.
  Other Names: Anodal transcranial direct current stimulation; Non invasive brain stimulation
  Arms: Real tDCS; Sham tDCS

SUMMARY:
This study evaluates the effects of corticosteroid injections over time, as well as the additional effect provided by subsequent transcranial direct current stimulation (tDCS) of the motor cortex on patients with rotator cuff tendinopathy of the shoulder. All patients will receive a subacromial corticosteroid injection. Two weeks later, a third will receive a treatment of tDCS, a third will receive a placebo a-tDCS treatment, and the last third will not receive any additional treatment.

DETAILED DESCRIPTION:
Corticosteroid injections (CSI) are often used by physicians in the treatment of rotator cuff tendinopathy, a painful chronic degeneration of the tendons in the shoulder. However, the effect of CSI in comparison with placebo is disputed in the scientific literature, with most studies only showing mild short-term effect (less than six weeks) on pain compared to placebo injections.

Transcranial direct current stimulation (tDCS) is a non-invasive technique allowing to stimulate areas of the brain in order to change the excitability of the neurons. When the negative electrode is applied on the motor cortex of the brain, it increases the excitability of the neurons in that area, which in turns inhibits the activity of the thalamus, an area of the brain linked with the perception of pain. Some studies have shown that tDCS can improve chronic pain of different origins, such as lower back pain, fibromyalgia, stroke, osteoarthritis, and post-operative pain.

We tested whether applying tDCS following a CSI would have more effect on patient's pain, function, and activity, than CSI alone.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder pain for at least 9 months
* Trial of conservative treatment prior to inclusion
* Positive painful arc sign
* At least one positive impingement test (Neer or Hawkin's impingement sign)
* Written and oral comprehension of French and/or English

Exclusion Criteria specific to rotator cuff tendinopathy and CSI:

* Traumatic origin
* Diagnosis of a systemic inflammatory joint disease
* Complete rotator cuff tear on physical examination or MRI
* Diagnosis of acromio-clavicular syndrome
* Presence of cervical nerve root pain or symptoms
* Other confounding pathologies seen clinically or radiographically
* History of previous fracture or surgery at the shoulder
* Contraindication to CSI
* CSI received in the last three months
* Planned or ongoing pregnancy
* Receiving worker's compensation or being involved in litigation relating to the shoulder pathology.
* Inability to follow protocol instructions

Exclusion Criteria specific to tDCS and transcranial magnetic stimulation:

* History of epilepsy or convulsions
* Brain metallic implants or fragments
* Brain lesions or tumors
* Use of a pacemaker or ICD
* Use of an intravenous medication pump
* Severe cardiac disease, or recent cardiac event
* Consumption of medications known to lower the seizure threshold
* Alcoholism
* Severe sleep deprivation
* Eczema or skin lesions at the area of electrode application

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2016-03-16 (Actual); Study Completion 2016-03-16 (Actual)

PRIMARY OUTCOMES:
Western Ontario Rotator Cuff index (WORC) | Two weeks following tDCS (four weeks after CSI)
  The WORC is a health related quality of life questionnaire developed specifically to assess outcome in patients with rotator cuff disease. It includes 21 questions in the form of visual analog scales (VAS) covering five domains: physical symptoms, sports and recreation, work, quality of life, and emotional status. The final score can be reported over 100 points, with a higher score represents better function.

SECONDARY OUTCOMES:
Western Ontario Rotator Cuff index (WORC) | One week before the CSI, day of the CSI (just prior to the injection), two-weeks after CSI (just prior to tDCS),eight weeks after CSI (six weeks after tDCS)
  The WORC is a health related quality of life questionnaire developed specifically to assess outcome in patients with rotator cuff disease. It includes 21 questions in the form of visual analog scales (VAS) covering five domains: physical symptoms, sports and recreation, work, quality of life, and emotional status. The final score can be reported over 100 points, with a higher score represents better function.
Short version of the Disability of the Arm, Shoulder and Hand questionnaire (QuickDASH) | One week before the CSI, day of the CSI (just prior to the injection), two-weeks after CSI (just prior to tDCS), four weeks after CSI, eight weeks after CSI
  The QuickDASH is a health related quality of life questionnaire developed for pathologies affecting the arm, shoulder and hand. It consists of 11 questions in the form of Likert scales. The score can be reported on a scale of 0 to 100, with higher score representing worse outcome.
Pain visual analog scale (pain VAS) | Filled every day, but it will be averaged for every week, starting one week before the CSI and ending four weeks after, with an additional week eight weeks following CSI.
  The participant will be asked to rank their pain for the last 24h on a VAS, with anchors being "no pain" on the left end, and "Extreme pain" on the right end.
Shoulder Range of Motion (ROM) | One week before the CSI, day of the CSI (just prior to the injection), two-weeks after CSI (just prior to tDCS), four weeks after CSI
  Shoulder ROM will be measured using a goniometer and reported in degrees in six different planes: abduction, flexion, scapular elevation (scaption), external rotation with the arm at the side, external rotation with the arm abducted 90 degrees and internal rotation with the arm abducted 90 degree.
  Additionally, internal rotation will also be measured visually with the maximal spinal level reached by the thumb with the hand at the back.
Shoulder strength | One week before the CSI, day of the CSI (just prior to the injection), two-weeks after CSI (just prior to tDCS), four weeks after CSI
  Using a hand-held dynamometer, shoulder strength will be measured in three planes: scapular plane with the thumb pointed down (Jobe test, or empty can test), external rotation with the arm adducted, internal rotation with the arm adducted
Shoulder activity VAS | Filled every day, but it will be averaged for every week, starting one week before the CSI and ending four weeks after, with an additional week eight weeks following CSI.
  The participants will be asked to rank their estimated affected shoulder use for the last 24h using a VAS, with the left anchor being "Not at all" and the right anchor being "All the time".
Arm usage measured by actimetry | Worn every day, but it will be averaged for every week, starting one week before the CSI and ending four weeks after.
  An accelerometer developed at our institution (WIMU-GPS) will be worn at the wrist during the day for a total of five weeks. It will record acceleration, angular velocity, and magnetic field interactions in order to estimate upper extremity usage. At the time of initial ethical approval, the exact algorithm for upper extremity usage estimation was not decided. At the end of data collection, it was decided to use percentage of active time (time spent over a prespecified threshold), activity count, ratio of high intensity activities (activities in the highest 33% percentile of activity count), ratio of medium intensity activities (activities in the middle 33% percentile of activities) and ratio of low intensity activities (activities in the low 33% percentile of activity counts)

OTHER OUTCOMES:
Global rating of change scale (GRCS) | Two week follow the CSI (prior to tDCS), four weeks following CSI (two weeks after tDCS), eight weeks after CSI (six weeks after tDCS).
  This form asks the participants to rate improvement in their symptoms on a scale with 15 levels, starting from "A very great deal worse", with a midpoint being "About the same" and ending with "A very great deal better". This questionnaire will be used to help validate accelerometry as an outcome measure in a secondary analysis.
Percentage of improvement | Two week follow the CSI (prior to tDCS), four weeks following CSI (two weeks after tDCS).
  Participants will be asked verbally how much improvement, in percentage, they felt their shoulder improved since the CSI.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Boissy, PhD, Study Director — Université de Sherbrooke

IPD SHARING:
Plan to Share IPD: Undecided
We will likely be sharing an spreadsheet containing anonymized IPD, including all outcome measures for each time point. The accelerometer data will however be summarized in a per-week average and standard deviation, as the data files are too large (>4 Gb each) to be shared in a practical way.
  We also plan to share original study protocol, analysis plan, and participant consent forms. The data will be available for a total of 5 years after publication of the study results, and then destroyed as required by our research ethics board.

REFERENCES:
- [Derived] Larrivee S, Balg F, Leonard G, Bedard S, Tousignant M, Boissy P. Transcranial direct current stimulation (a-tCDS) after subacromial injections in patients with subacromial pain syndrome: a randomized controlled pilot study. BMC Musculoskelet Disord. 2021 Mar 11;22(1):265. doi: 10.1186/s12891-021-04139-2. PMID 33706729

DOCUMENTS (1):
  • Informed Consent Form (2015-02-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT03967574/ICF_000.pdf